CLINICAL TRIAL: NCT05245955
Title: Feasibility and Validity of Robotic Assessments With the ReHapticKnob to Characterize Kinaesthesia and Haptic Perception of the Hand in Patients With Parkinson's Disease: an Exploratory Study
Brief Title: Robotic Assessments of Hand Function in Patients With Parkinson's Disease
Acronym: RHK Parkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Clinica Hildebrand Brissago (Other); Neurocentro - Istituto di Neuroscienze Cliniche della Svizzera Italiana (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHK Parkinson
Record Dates: First submitted 2021-11-11; First posted 2022-02-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Sensory impairments; Kinaesthesia; Haptic perception; Robot-assisted assessments; Assessment of the hand sensory function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic assessment of sensory hand function (Experimental): This arm involves a group of persons with Parkinson's disease and an age-matched control group. Both groups undergo the assessments of kinaesthesia and haptic perception of the hand implemented on the ReHapticKnob.
  Interventions: Device: Assessments of the hand sensory function with the ReHapticKnob

INTERVENTIONS:
Device: Assessments of the hand sensory function with the ReHapticKnob — During the assessment sessions with the ReHapticKnob, subjects sit comfortably on a chair in front of a screen and place the fingers of the hand on the handles of the device. The different assessments consist of moving the hand or forearm of the subjects to two different positions and asking the subject to discriminate between them (discrimination thresholds for the amplitude of grasping and forearm pronosupination positions), of passively moving the hand or forearm of the subject at low velocities and asking the subject to say when he/she detects the movement (detection thresholds for passive movements), or of rendering two objects with different stiffness and asking the subject to discriminate between them (discrimination thresholds for the stiffness of objects pinched with the hand).

SUMMARY:
It has been shown that patients with Parkinson's disease (PD) have impaired kinaesthesia and haptic perception of the upper limbs. In PD patients, these impairments might be involved in the development of hypometria or bradykinesia and may play a role in postural deficits, thereby significantly contributing to the overall disability level.

Dedicated conventional or robot-assisted training might improve sensory-motor function in PD patients. In order to provide efficient robot-assisted therapy, robotic devices have to be able to tailor the therapy difficulty to the individual impairment profile of each patient. For difficulty adaptation in robot-assisted therapy, it is important to assess the impairment profiles with the same robotic platform that would be used for therapy, therefore minimizing costs or potential errors coming from the use of different devices. However, up to now, little emphasis has been placed on providing sensory-motor robot-assisted therapy for the upper limbs to persons with PD based on their individual level of impairment.

The aim of this study is therefore to evaluate if the assessments of sensory-motor hand function implemented on a robotic device for hand rehabilitation, i.e. the ReHapticKnob, are suitable to measure the impairments of kinaesthesia and haptic perception observed in subjects with Parkinson's disease.

If the assessments implemented in the ReHapticKnob are sensitive enough to detect a difference between the sensory-motor function of PD patients and healthy subjects, the device might in the future be used to assess improvements before and after sensory-motor therapy. This is a necessary step before the investigators can use these assessments to tailor the difficulty level of the therapy performed with the ReHapticKnob and to investigate the benefits and impact of such a therapy on the kinaesthetic and haptic impairments of persons with PD.

ELIGIBILITY:
Ten patients with Parkinson's disease and 10 age-matched control subjects will be recruited.

Patients with Parkinson's disease: inclusion criteria

* Diagnosis of idiopathic Parkinson's disease according to UK Parkinson's disease society brain bank clinical diagnostic criteria
* Age between 35 and 80 years
* Hoehn and Yahr stage of I, II or III during the ON state
* Montreal Cognitive Assessment (MoCA) ≥ 26
* No tremor, i.e.:

  * Postural tremor for the hand: MDS-UPDRS 3.15 < 1
  * Kinetic tremor of the hands: MDS-UPDRS 3.16 ≤ 1
  * Rest tremor amplitude for the extremities: MDS-UPDRS 3.17 < 1
  * Constancy of rest tremor: MDS-UPDRS 3.18 < 1
* The subject read, understood and signed the informed consent

Patients with Parkinson's disease: exclusion criteria

* Polyneuropathy registered in the anamnesis or peripheral sensory-motor impairments detected in a neurological clinical examination
* Mild to severe dyskinesia of the upper limbs: point 5 of the Abnormal Involuntary Movement Scale (AIMS) > 1
* Orthopedic pathologies of the upper limbs or other pathologies possibly interfering with the study
* Pacemaker, deep-brain-stimulator or other active implanted devices

Control subjects: inclusion criteria

* Age between 35 and 80 years
* Montreal Cognitive Assessment (MoCA) ≥ 26
* The subject read, understood and signed the informed consent

Control subjects: exclusion criteria

* Any history of neurological, orthopaedic or rheumatologic disease affecting the upper limbs or other pathologies possibly interfering with the study
* Pacemaker or other active implanted devices

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Detection threshold resulting from the assessment of detection of passive grasping movements - Right hand | Through study completion, an average of 2 weeks
  Outcome of the assessment for the detection of passive grasping movements performed with the right hand. This threshold is expressed in time until movement detection.
Detection threshold resulting from the assessment of detection of passive grasping movements - Left hand | Through study completion, an average of 2 weeks
  Outcome of the assessment for the detection of passive grasping movements performed with the left hand. This threshold is expressed in time until movement detection.
Detection threshold resulting from the assessment of detection of passive forearm pronosupination movements - Right forearm | Through study completion, an average of 2 weeks
  Outcome of the assessment for the detection of passive forearm pronosupination movements performed with the right forearm. This threshold is expressed in time until movement detection.
Detection threshold resulting from the assessment of detection of passive forearm pronosupination movements - Left forearm | Through study completion, an average of 2 weeks
  Outcome of the assessment for the detection of passive forearm pronosupination movements performed with the left forearm. This threshold is expressed in time until movement detection.
Discrimination threshold resulting from the assessment of just noticeable difference for grasping positions - Right hand | Through study completion, an average of 2 weeks
  Outcome of the assessment for the discrimination of grasping positions performed with the right hand. This threshold is expressed in millimeters and represents the minimum difference that the subject can perceive.
Discrimination threshold resulting from the assessment of just noticeable difference for grasping positions - Left hand | Through study completion, an average of 2 weeks
  Outcome of the assessment for the discrimination of grasping positions performed with the left hand. This threshold is expressed in millimeters and represents the minimum difference that the subject can perceive.
Discrimination threshold resulting from the assessment of just noticeable difference for pronosupination positions - Right forearm | Through study completion, an average of 2 weeks
  Outcome of the assessment for the discrimination of pronosupination positions performed with the right forearm. This threshold is expressed in degrees and represents the minimum difference that the subject can perceive.
Discrimination threshold resulting from the assessment of just noticeable difference for pronosupination positions - Left forearm | Through study completion, an average of 2 weeks
  Outcome of the assessment for the discrimination of pronosupination positions performed with the left forearm. This threshold is expressed in degrees and represents the minimum difference that the subject can perceive.
Discrimination threshold resulting from the assessment of haptic perception - Right hand | Through study completion, an average of 2 weeks
  Outcome of the assessment for haptic perception performed with the right hand. This threshold is expressed as Weber Fraction and represents the minimum difference in stiffness that the subject can perceive.
Discrimination threshold resulting from the assessment of haptic perception - Left hand | Through study completion, an average of 2 weeks
  Outcome of the assessment for haptic perception performed with the left hand. This threshold is expressed as Weber Fraction and represents the minimum difference in stiffness that the subject can perceive.

SECONDARY OUTCOMES:
Demographic information | This information is collected during the screening visit performed at the beginning of the study (day 0).
  Gender, age, year of birth.
Edinburgh Handedness Inventory Score | This information is collected during the screening visit performed at the beginning of the study (day 0).This information is collected during the screening visit performed at the beginning of the study (day 0).
  Questionnaire to define handedness.
Montreal Cognitive Assessment | This information is collected during the screening visit performed at the beginning of the study (day 0).This information is collected during the screening visit performed at the beginning of the study (day 0).
  Assessment of cognitive function (max score = 30, high score = better).
Proprioception item of the Nottingham Sensory Assessment | The control group does this assessment during the screening visit (day 0). The group of patients with Parkinson's disease does this during the second examination visit (day 0 to day 0 + 2 days).
  Assessments used to characterize proprioception.
MDS-Unified Parkinson's Disease Rating Scale: items 3.15 to 3.18 | This information is collected during the screening visit performed at the beginning of the study (day 0).
  Scale to characterize the state of the Parkinson's disease. This is done for the group of patients with Parkinson's disease only. These items are performed at the beginning as they are considered for the inclusion criteria.
MDS-Unified Parkinson's Disease Rating Scale III | This information is collected during the second examination visit (day 0 to day 0 + 2 days).
  Scale to characterize the state of the Parkinson's disease. This is done for the group of patients with Parkinson's disease only.
Hoehn and Yahr stage | This information is collected during the screening visit performed at the beginning of the study (day 0).
  Scale to characterize the state of the Parkinson's disease. This is done for the group of patients with Parkinson's disease only.
Abnormal Involuntary Movement Scale | This information is collected during the screening visit performed at the beginning of the study (day 0).
  Scale to characterize the state of the Parkinson's disease. This is done for the group of patients with Parkinson's disease only.
Levodopa equivalent daily dose | This information is collected during the second examination visit (day 0 to day 0 + 2 days).
  Information used to characterize the state of the Parkinson's disease and the timespan when the patient is in the ON state. This is collected for the group of patients with Parkinson's disease only.
Disease onset | This information is collected during the second examination visit (day 0 to day 0 + 2 days).
  Information used to characterize the state of the Parkinson's disease. This is collected for the group of patients with Parkinson's disease only.
Most affected side | This information is collected during the second examination visit (day 0 to day 0 + 2 days).
  Information used to characterize the side of the body most affected by the Parkinson's disease. This is collected for the group of patients with Parkinson's disease only.
Frontal Assessment Battery | This assessment is performed once during the study (from day 0 to day 0 + 25 days).
  Assessment of cognitive function. This is collected for the group of patients with Parkinson's disease only.
Attentive matrices | This assessment is performed once during the study (from day 0 to day 0 + 25 days).
  Assessment of cognitive function. This is collected for the group of patients with Parkinson's disease only.
Digit span | This assessment is performed once during the study (from day 0 to day 0 + 25 days).
  Assessment of cognitive function. This is collected for the group of patients with Parkinson's disease only.
Fatigue scale for motor and cognitive functions | This assessment is performed once during the study (from day 0 to day 0 + 25 days).
  Assessment of cognitive function. This is collected for the group of patients with Parkinson's disease only.

CONTACTS AND LOCATIONS:
Overall Officials: Daria Dinacci, Dr. med., Principal Investigator — Clinica Hildebrand Centro di riabiliazione Brissago
Locations (1):
- Clinica Hildebrand, Centro di Rehabilitazione Brissago, Brissago, Switzerland

IPD SHARING:
Plan to Share IPD: No